CLINICAL TRIAL: NCT03597945
Title: Magnesium-sulfate as Adjuvant in Prehospital Femoral Nerve Block for Patient With Diaphysial Femoral Fracture: a Randomized Controlled Trial
Brief Title: Magnesium-sulfate as Adjuvant in Prehospital Femoral Nerve Block for Patient With Diaphysial Femoral Fracture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Mohamed Kahloul, principal investigator, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS 1842015
Record Dates: First submitted 2018-06-25; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Acute Pain Due to Trauma
Keywords: Magnesium sulfate; lidocaine; femoral nerve block; prehospital; pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Epinephrine; Saline Solution; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of two groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Placebo (Placebo Comparator): For patients of this group, the intervention was a femoral nerve block with:
  * 15 ml of lidocaine with epinephrine (300 mg)
  * and 3 ml of normal saline as adjuvant.
  Interventions: Procedure: lidocaine with epinephrine; Procedure: normal saline
- Group Magnesium (Active Comparator): For patients of this group, the intervention was a femoral nerve block with:
  * 15 ml of lidocaine with epinephrine (300 mg)
  * and 3 ml of Magnesium sulfate 15% (450 mg) as adjuvant.
  Interventions: Procedure: lidocaine with epinephrine; Procedure: Magnesium sulfate

INTERVENTIONS:
Procedure: lidocaine with epinephrine — lidocaine with epinephrine in prehospital femoral nerve block for patient with diaphysial femoral fracture
Procedure: normal saline — normal saline as adjuvant to lidocaine with epinephrine in prehospital femoral nerve block for patient with diaphysial femoral fracture
  Arms: Group Placebo
Procedure: Magnesium sulfate — Magnesium-sulfate as adjuvant to lidocaine with epinephrine in prehospital femoral nerve block for patient with diaphysial femoral fracture
  Arms: Group Magnesium

SUMMARY:
Prehospital management of traumatic pain is commonly based on morphine while loco-regional analgesia techniques, especially the femoral nerve block (FNB), can be safely and efficiently used. Adjuvants uses can reduce local anesthetic doses and decrease their related risk. The aim of the study was to assess the analgesic effect of Magnesium sulfate (Mg S) when used as adjuvant in prehospital FNB.

This is a randomized double-blinded trial conducted in a prehospital medical department of an academic hospital. Patients with isolated diaphysial femoral fracture and eligible to participate were randomized into 2 groups. The Group Placebo had a FNB with 15 ml of lidocaine with epinephrine (300 mg) and 3 ml of normal saline. The Group Magnesium had a FNB with 15 ml of lidocaine with epinephrine (300 mg) and 3 ml of Mg S 15% (450 mg). The FNB was performed according to the WINNIE technique. Primary endpoints were morphine consumption and pain intensity during the first 6 hours. Secondary end-points were the duration of the sensitive block, time to the first analgesic request, side effects occurrence.

DETAILED DESCRIPTION:
After approval by the Research Ethics Board, this randomized double-blinded clinical trial was carried out in the prehospital medical department of a Tunisian teaching hospital over a 3 years period (April 30, 2015 to April 29, 2018). All patients with isolated diaphysial femoral fracture were enrolled. Inclusion criteria were age over 18 years, informed and writing consent.

Based on the results of a previous study and targeting a decrease of 1 cm in pain intensity assessed by the visual analogue score (VAS), the sample size was assessed to be at least 22 patients in each study group, considering a threshold of 0.05 and a study power of 90%. Sample size was increased in each group to 25 patients to allow possible dropouts.

Included patients randomly received, in a double-blind manner (using computer-generated allocation numbers sealed in brown envelopes), one of two local anesthetic solutions.

The control group (Group Placebo) had a FNB with 15 ml of lidocaine with epinephrine 0,005 mg/ml (300 mg) and 3 ml of normal saline.

The intervention group (Group Magnesium) had a FNB with 15 ml of lidocaine with epinephrine 0,005 mg/ml (300 mg) and 3 ml of Mg S 15% (450 mg).

FNB was performed according to WINNIE technique after rigorous asepsis. Its efficiency was evaluated 15 minutes after by pinprick test. Pain was assessed by visual analog scale (VAS) every 10 minutes for the first hour, then every 60 minutes until the 6th hour after the block. Patients with a VAS > 3 received morphine titration.

Primary endpoints were morphine consumption and pain intensity during the first 6 hours.

Secondary end-points were the duration of the sensitive block, time to the first analgesic request, the occurrence of side effects (erythematic, sedation, decrease in average blood pressure, or heart rate of more than 15% of the initial basic value).

ELIGIBILITY:
Inclusion Criteria:

* patients with isolated diaphysial femoral fracture
* age over 18 years
* informed and writing consent

Exclusion Criteria:

* body mass index over 30
* fracture associated with vascular or sensory disorders
* cardiovascular diseases
* hepatic or renal impairments
* neuromuscular diseases
* opioids administration before the FNB
* chronic pain
* a long-term pain relief treatment
* pretreatment with calcium or calcium antagonist
* known allergy to one of the study drugs
* infection at the injection site
* open fracture
* fracture undocumented by the imagery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2018-04-29 (Actual)

PRIMARY OUTCOMES:
morphine consumption | first 6 hours
  morphine requirements during the first 6 hours (mg)
pain intensity: visual analog scale (VAS) | first 12 hours
  pain intensity during the first 6 hours assessed by the visual analog scale (VAS)

SECONDARY OUTCOMES:
sensitive block duration | first 6 hours
  the duration of the sensitive block (in minutes)
time to the first analgesic request | first 6 hours
  time to the first analgesic request in minutes
side effects occurrence | first 12 hours
  the occurrence of side effects such as erythematic, sedation, decrease in average blood pressure, or heart rate of more than 15% of the initial basic value.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Kahloul, MD, Principal Investigator — Faculty of Medicine, Sousse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fawcett WJ, Haxby EJ, Male DA. Magnesium: physiology and pharmacology. Br J Anaesth. 1999 Aug;83(2):302-20. doi: 10.1093/bja/83.2.302. PMID 10618948
- [Result] Capdevila X, Biboulet P, Bouregba M, Rubenovitch J, Jaber S. Bilateral continuous 3-in-1 nerve blockade for postoperative pain relief after bilateral femoral shaft surgery. J Clin Anesth. 1998 Nov;10(7):606-9. doi: 10.1016/s0952-8180(98)00097-x. PMID 9805704
- [Result] Schiferer A, Gore C, Gorove L, Lang T, Steinlechner B, Zimpfer M, Kober A. A randomized controlled trial of femoral nerve blockade administered preclinically for pain relief in femoral trauma. Anesth Analg. 2007 Dec;105(6):1852-4, table of contents. doi: 10.1213/01.ane.0000287676.39323.9e. PMID 18042893
- [Result] Mukherjee K, Das A, Basunia SR, Dutta S, Mandal P, Mukherjee A. Evaluation of Magnesium as an adjuvant in Ropivacaine-induced supraclavicular brachial plexus block: A prospective, double-blinded randomized controlled study. J Res Pharm Pract. 2014 Oct;3(4):123-9. doi: 10.4103/2279-042X.145387. PMID 25535620
- [Result] Bondok RS, Abd El-Hady AM. Intra-articular magnesium is effective for postoperative analgesia in arthroscopic knee surgery. Br J Anaesth. 2006 Sep;97(3):389-92. doi: 10.1093/bja/ael176. Epub 2006 Jul 11. PMID 16835255
- [Derived] Jebali C, Kahloul M, Hassine N, Jaouadi MA, Ferhi F, Naija W, Chebili N. Magnesium Sulfate as Adjuvant in Prehospital Femoral Nerve Block for a Patient with Diaphysial Femoral Fracture: A Randomized Controlled Trial. Pain Res Manag. 2018 Dec 3;2018:2926404. doi: 10.1155/2018/2926404. eCollection 2018. PMID 30631386